CLINICAL TRIAL: NCT01977547
Title: Age of Blood in Children in Pediatric Intensive Care Units
Acronym: ABC-PICU
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Canadian Institutes of Health Research (CIHR) (Other Government); Ministere de la Sante et des Services Sociaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201302030; 1U01HL116383-01 (NIH); MOP 126113 (Other Grant/Funding Number: Canadian Institutes of Health Research (CIHR))
Record Dates: First submitted 2013-08-09; First posted 2013-11-06 (Estimated); Results first posted 2021-04-29 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Anemia
Keywords: Red blood cell transfusions; Red blood cell storage age; Pediatrics; Critical Care
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Short storage (Active Comparator): Red blood cells storage duration of equal to or less than 7 days.
  Interventions: Biological: Short storage RBC age
- Standard issue (Active Comparator): Red blood cells storage duration of 2 to 42 days with an expected average length of storage of about 17-21 days.
  Interventions: Biological: Short storage RBC age

INTERVENTIONS:
Biological: Short storage RBC age — IND obtained to cover the expiration date on the red blood cell unit

SUMMARY:
ABC PICU is a randomized clinical trial that will compare the clinical consequences of RBC storage duration in 1538 critically ill children. Laboratory and observational evidence points to serious concerns about the lack of safety and effectiveness of older RBCs, especially in more vulnerable populations. Physicians and institutions have been systematically transfusing fresh RBCs to some pediatric patients primarily because of beliefs that the use of fresh RBCs improve outcomes. Conversely, the standard practice of blood banks is to deliver the oldest RBC unit in order to decrease blood wastage. To provide much needed high quality evidence to answer the question "do RBCs of reduced storage duration improve outcomes?" The ABC PICU Trial will conduct a RCT comparing development of New or Progressive Multiple Organ Dysfunction Syndrome (NPMODS) in critically ill children transfused with either RBCs stored ≤ 7 days or standard issue RBCs (expected mean RBC storage duration of 17-21 days).

ELIGIBILITY:
Patients are considered eligible to participate in the trial if one of the following occur:

1. First RBC transfusion is requested within the first 7 days (168 hours) of ICU admission.

   OR
2. First RBC transfusion is requested for a patient in the Emergency Room, and the PICU team is involved with the clinical care of the patient, and the patient will definitively be transferred to the ICU.

   OR
3. Patient assessed pre-operatively and for whom ICU admission is planned post-operatively, and who is determined to definitively require a first RBC transfusion during surgery.

Inclusion Criteria:

Eligible critically ill pediatric patients who have an expected length of stay after transfusion in the ICU > 24 hours based on the best judgment of the attending ICU staff.

Exclusion Criteria:

* Age at time of enrollment < 3 days from birth or has reached their 16th birthday.
* Post-conception age < 36 weeks at time of enrollment
* Documented RBC transfusion within the 28 days prior to fulfilling the eligibility criteria
* Previously randomized in this study
* Weight < 3.0 kg on ICU admission
* Known Pregnancy
* Conscious objection or unwillingness to receive blood products
* Not expected to survive beyond 24 hours, brain death or suspected brain death
* Limitation or withdrawal of care decisions have been made
* Enrollment in another randomized clinical trial which has not been approved for co-enrollment
* Patients for whom autologous and/or directed donation RBCs will be provided
* Patients for whom the treating physician routinely and systematically requests RBC ≤ 14 days of storage
* Patients for whom there systematically exist RBC aliquoting policies that mandate the initial use of units stored ≤ 14 days (ex: Pedi-Pack).
* On ECMO or plan to be immediately placed on ECMO at time of enrollment
* Patient predicted or presumed to require a massive transfusion (> 40ml/kg of all blood components in a 24 hour period) according to treating physician judgment
* Refusal by physician
* Inability to obtain consent
* Blood bank personnel experiences difficulties in securing blood products (difficult cross matches, rare blood groups and diseases like IgA deficiency)
* Insufficient number of ABO type compatible RBC units available in the blood bank at randomization with a storage time ≤ 7 days (minimum 1 unit regardless of patient age)
* All RBC units available for the patient are not leukocyte-reduced prior to storage

Ages: 3 Days to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1538 (Actual)
Dates: Start 2014-01; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip C. Spinella, MD, Principal Investigator — Washington University School of Medicine, St. Louis; Marisa Tucci, MD, Principal Investigator — Ste-Justine Hospital, Montreal
Locations (37):
- United States (20):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Diamond Children's Medical Center, Tucson, Arizona
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - University of California, San Francisco, San Francisco, California
  - The Children's Hospital and University of Colorado Denver School of Medicine, Aurora, Colorado
  - UF Health Shands Children's Hospital, Gainesville, Florida
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Lutheran General Hospital, Park Ridge, Illinois
  - James Whitcomb Riley Hospital for Children, Indianapolis, Indiana
  - Washington University School of Medicine, St Louis, Missouri
  - Weill Cornell Medical College, New York, New York
  - Golisano Children's Hospital at Strong, Rochester, New York
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Medical Center Dallas, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Canada (7):
  - Stollery Children's Hospital, Edmonton, Alberta
  - IWK Health Centre, Halifax, Nova Scotia
  - London Health Sciences Centre, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - CHU Sainte Justine, Montreal, Quebec
  - Centre Hospitalier de I'Universite Laval, Québec
- France (7):
  - Hôpital Necker-enfants, Paris, Malades Paris
  - Place Amélie Raba Léon, Bordeaux
  - Hôpital Jeanne de Flandre, Lille
  - Hôpital Mère Enfant, Nantes
  - Hôpital Robert Debré, Paris
  - Hôpital Universitaire Necker - Enfants Malades, Paris
  - CHU Pontchaillou, Rennes
- Sheba Medical Center, Tel Litwinsky, Israel
- Italy (2):
  - Meyer's Hospital, Florence
  - Bamino Gesú, Rome

REFERENCES:
- [Derived] Spinella PC, Tucci M, Fergusson DA, Lacroix J, Hebert PC, Leteurtre S, Schechtman KB, Doctor A, Berg RA, Bockelmann T, Caro JJ, Chiusolo F, Clayton L, Cholette JM, Guerra GG, Josephson CD, Menon K, Muszynski JA, Nellis ME, Sarpal A, Schafer S, Steiner ME, Turgeon AF; ABC-PICU Investigators, the Canadian Critical Care Trials Group, the Pediatric Acute Lung Injury and Sepsis Investigators Network, the BloodNet Pediatric Critical Care Blood Research Network, and the Groupe Francophone de Reanimation et Urgences P. Effect of Fresh vs Standard-issue Red Blood Cell Transfusions on Multiple Organ Dysfunction Syndrome in Critically Ill Pediatric Patients: A Randomized Clinical Trial. JAMA. 2019 Dec 10;322(22):2179-2190. doi: 10.1001/jama.2019.17478. PMID 31821429
- [Derived] Tucci M, Lacroix J, Fergusson D, Doctor A, Hebert P, Berg RA, Caro J, Josephson CD, Leteurtre S, Menon K, Schechtman K, Steiner ME, Turgeon AF, Clayton L, Bockelmann T, Spinella PC; Canadian Critical Care Trials Group; Pediatric Critical Care Blood Research Network (BloodNet); Pediatric Acute Lung Injury and Sepsis Investigators (PALISI) Network. The age of blood in pediatric intensive care units (ABC PICU): study protocol for a randomized controlled trial. Trials. 2018 Jul 28;19(1):404. doi: 10.1186/s13063-018-2809-y. PMID 30055634

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Short Storage | Standard Issue
Started | 768 | 770
Completed | 728 | 733
Not Completed | 40 | 37

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Short Storage | Standard Issue | Total
Number analyzed (Participants) | 728 | 733 | 1461
Age, Continuous [Median (Inter-Quartile Range); unit: year] | 1.8 [0.5 to 6.9] | 1.9 [0.5 to 7.0] | 1.8 [0.5 to 7.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 352 | 339 | 691
  Male | 376 | 394 | 770
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 68 | 82 | 150
  Not Hispanic or Latino | 515 | 508 | 1023
  Unknown or Not Reported | 145 | 143 | 288
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 22 | 11 | 33
  Asian | 37 | 29 | 66
  Native Hawaiian or Other Pacific Islander | 5 | 4 | 9
  Black or African American | 86 | 103 | 189
  White | 399 | 415 | 814
  More than one race | 24 | 13 | 37
  Unknown or Not Reported | 155 | 158 | 313
Region of Enrollment [Number; unit: participants]
  Canada | 196 | 194 | 390
  United States | 415 | 423 | 838
  Italy | 19 | 18 | 37
  Israel | 6 | 9 | 15
  France | 92 | 89 | 181

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With New or Progressive Multiple Organ Dysfunction Syndrome (NPMODS)
Description: The primary outcome measure of this RCT is NPMODS defined as the proportion of patients who die during the 28 days after randomization or who develop NPMODS. For patients with no organ dysfunction at randomization, New MODS is the development of ≥ 2 concurrent organ dysfunctions during the 28 days after randomization. For patients with 1 organ dysfunction at randomization, New MODS is the development of at least 1 other concurrent organ dysfunction after randomization. Patients with MODS (ie concurrent dysfunction of ≥ 2 organ systems) at randomization can develop Progressive MODS defined as development of at least 1 additional concurrent organ dysfunction at during the 28 days after randomization. All deaths will be considered Progressive MODS. NPMODS will be monitored up to 28 days or ICU discharge because it is almost never observed beyond this time in children.
Time Frame: 28 days after randomization
Population: Development of organ dysfunction in all participants
Measure: Count of Participants; unit: Participants
Arm/Group | Short Storage | Standard Issue
Number analyzed (Participants) | 728 | 732
Participants | 147 | 133

2. Secondary Outcome: Organ Dysfunction
Description: Difference in number of organ dysfunctions.
Time Frame: Up to 28 days after randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Short Storage | Standard Issue
Number analyzed (Participants) | 669 | 732
Participants | 129 | 133

3. Secondary Outcome: PELOD-2 Score
Description: Difference in PELOD-2 score. Change from randomization to Worst PELOD-2 score. (Pediatric Logistic Organ Dysfunction) Points are on a range of 0-6 and based on Neurologic, cardiovascular, renal, respiratory, and hematologic function. The higher the score the worse the organ failure is and higher mortality rate.
Time Frame: Up to 28 days after randomization.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Short Storage | Standard Issue
Number analyzed (Participants) | 728 | 733
score on a scale | 0.5 (5.8) | -0.05 (4.7)

4. Secondary Outcome: Nosocomial Infection
Description: Difference in nosocomial infection rate.
Time Frame: Up to 28 days after randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Short Storage | Standard Issue
Number analyzed (Participants) | 728 | 732
Participants | 24 | 23

5. Secondary Outcome: Sepsis, Severe Sepsis, Septic Shock
Description: Difference in the rate of sepsis, severe sepsis or septic shock.
Time Frame: Up to 28 days after randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Short Storage | Standard Issue
Number analyzed (Participants) | 619 | 608
Participants
  Sepsis | 160 | 154
  Severe Sepsis | 63 | 60
  Septic Shock | 59 | 57

6. Secondary Outcome: Acute Respiratory Distress Syndrome
Description: Difference in the rate of acute respiratory distress syndrome.
Time Frame: Up to 28 days after randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Short Storage | Standard Issue
Number analyzed (Participants) | 619 | 608
Participants | 41 | 29

7. Secondary Outcome: Mechanical Ventilation
Description: 28 day mechanical ventilation free days
Time Frame: Up to 28 days after randomization.
Measure: Mean (Inter-Quartile Range); unit: days
Arm/Group | Short Storage | Standard Issue
Number analyzed (Participants) | 728 | 733
days | 25.4 [19.6 to 27.9] | 25.8 [20.2 to 28.0]

8. Secondary Outcome: ICU Free Days
Description: Difference in ICU free days.
Time Frame: Up to 28 days after randomization
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Short Storage | Standard Issue
Number analyzed (Participants) | 728 | 733
days | 21.9 [14.5 to 25.3] | 22.0 [16.1 to 25.6]

9. Secondary Outcome: Mortality
Description: Difference in 90 day mortality.
Time Frame: Up to 90 days after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Short Storage | Standard Issue
Number analyzed (Participants) | 716 | 714
Participants | 49 | 45

10. Secondary Outcome: Delirium
Description: Transfusion Associated Delirium in pediatric critically ill children
Time Frame: up to 72 hours post last study transfusion
Measure: Count of Participants; unit: Participants
Arm/Group | Short Storage | Standard Issue
Number analyzed (Participants) | 69 | 77
Participants | 55 | 54

ADVERSE EVENTS:
Time Frame: 28 days for Adverse Events 90 days for mortality
Description: There is a change in the number of patients evaluated due to being lost to follow up in certain events.
Arm/Group | Short Storage | Standard Issue
All-Cause Mortality (participants affected / at risk) | 49/716 | 45/714
Serious Adverse Events (participants affected / at risk) | 80/728 | 84/733
Other Adverse Events (participants affected / at risk) | 0/728 | 0/733
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Short Storage (N=728) | Standard Issue (N=733)
Deep Vein Thrombosis (Blood and lymphatic system disorders) | 20 | 14
Hemolytic Transfusion Reaction (Blood and lymphatic system disorders) | 0 | 1
Hyperkalemia (Blood and lymphatic system disorders) | 30 | 36
Hypocalemia (Blood and lymphatic system disorders) | 10 | 13
Major Allergic Reaction (Immune system disorders) | 2 | 2
Nosocomial Pneumonia (Respiratory, thoracic and mediastinal disorders) | 18 | 15
Transfusion Associated Cardiac Overload (Blood and lymphatic system disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-13): https://cdn.clinicaltrials.gov/large-docs/47/NCT01977547/Prot_SAP_000.pdf